CLINICAL TRIAL: NCT05005910
Title: Efficacy of Vonoprazan Versus Intravenous Proton Pump Inhibitors for Prevention of Rebleeding in High Risk Peptic Ulcers Bleeding After Successful Endoscopic Hemostasis
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Uayporn Kaosombatwattana (Other)
Responsible Party: Sponsor-Investigator, Uayporn Kaosombatwattana, Lecturer, Mahidol University
Organization: Mahidol University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 011/2563
Record Dates: First submitted 2020-12-12; First posted 2021-08-16 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Peptic Ulcer With Haemorrhage
MeSH Terms: conditions — Peptic Ulcer Hemorrhage | interventions — 1-(5-(2-fluorophenyl)-1-(pyridin-3-ylsulfonyl)-1H-pyrrol-3-yl)-N-methylmethanamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vonoprazan (Experimental): Vonoprazan 20 mg oral every 12 hours (total 72 hours) then vonoprazan 20 mg oral once daily for 28 days
  Interventions: Drug: Vonoprazan
- PPIs (Active Comparator): PPIs IV infusion for 72 hours then oral PPIs twice per day for 28 days
  Interventions: Drug: PPIs IV infusion

INTERVENTIONS:
Drug: Vonoprazan — Vonoprazan 20 mg oral every 12 hours (total 72 hours)
  Arms: Vonoprazan
Drug: PPIs IV infusion — Pantoprazole 80 mg IV loading then 8 mg/hr
  Arms: PPIs

SUMMARY:
Upper gastrointestinal hemorrhage (UGIH) is common urgency condition.The estimate mortality rate about 7 percent from peptic ulcers disease(PUD). A proton pump inhibitors (PPIs) intravenous infusion are standard treatment for high risk ulcer bleeding. Vonoprazan,subclass of potassium-competitive acid blockers (P-CABs), have beneficial effects including rapid, long-lasting and strong acid suppression.The investigators design a randomized-controlled trial comparison between 72 hours of intravenous PPIs infusion and oral vonoprazan in high risk ulcer UGIH after achieve endoscopic hemostasis. Outcome measurement are re-bleeding rate in 30 days as primary and re-bleeding rate in 3 days, 30 days mortality, rate of angioembolisation, unit of blood transfusion, hospital cost and length of stay as secondary outcome.

ELIGIBILITY:
Inclusion Criteria:

* High risk peptic ulcers bleeding (Forrest class Ia,Ib,IIa,IIb)

Exclusion Criteria:

* Patients were not achieve endoscopic hemostasis
* End stage cancer disease
* Severe critical illness and ICU setting
* Uncorrectable coagulopathy
* Pregnancy or breast feeding
* Allergy to PPIs or Vonoprazan

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Rebleeding rate | 30 days

SECONDARY OUTCOMES:
Rebleeding rate | 3 days
Mortality rate | 30 days
Number of blood transfusion unit | 30 days
Rate of immobilisation or surgery | 30 days
Length of stay | Until discharge, assessed up to 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of internal medicine siriraj hospital, Mahidol university, Bangkok Noi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sung JJ, Suen BY, Wu JC, Lau JY, Ching JY, Lee VW, Chiu PW, Tsoi KK, Chan FK. Effects of intravenous and oral esomeprazole in the prevention of recurrent bleeding from peptic ulcers after endoscopic therapy. Am J Gastroenterol. 2014 Jul;109(7):1005-10. doi: 10.1038/ajg.2014.105. Epub 2014 Apr 29. PMID 24777150
- [Background] Tsoi KK, Hirai HW, Sung JJ. Meta-analysis: comparison of oral vs. intravenous proton pump inhibitors in patients with peptic ulcer bleeding. Aliment Pharmacol Ther. 2013 Oct;38(7):721-8. doi: 10.1111/apt.12441. Epub 2013 Aug 5. PMID 23915096
- [Background] Oshima T, Miwa H. Potent Potassium-competitive Acid Blockers: A New Era for the Treatment of Acid-related Diseases. J Neurogastroenterol Motil. 2018 Jul 30;24(3):334-344. doi: 10.5056/jnm18029. PMID 29739175
- [Background] Kagami T, Sahara S, Ichikawa H, Uotani T, Yamade M, Sugimoto M, Hamaya Y, Iwaizumi M, Osawa S, Sugimoto K, Miyajima H, Furuta T. Potent acid inhibition by vonoprazan in comparison with esomeprazole, with reference to CYP2C19 genotype. Aliment Pharmacol Ther. 2016 May;43(10):1048-59. doi: 10.1111/apt.13588. Epub 2016 Mar 18. PMID 26991399
- [Background] Miwa H, Uedo N, Watari J, Mori Y, Sakurai Y, Takanami Y, Nishimura A, Tatsumi T, Sakaki N. Randomised clinical trial: efficacy and safety of vonoprazan vs. lansoprazole in patients with gastric or duodenal ulcers - results from two phase 3, non-inferiority randomised controlled trials. Aliment Pharmacol Ther. 2017 Jan;45(2):240-252. doi: 10.1111/apt.13876. Epub 2016 Nov 27. PMID 27891632
- [Background] Sugano K, Kontani T, Katsuo S, Takei Y, Sakaki N, Ashida K, Mizokami Y, Asaka M, Matsui S, Kanto T, Soen S, Takeuchi T, Hiraishi H, Hiramatsu N. Lansoprazole for secondary prevention of gastric or duodenal ulcers associated with long-term non-steroidal anti-inflammatory drug (NSAID) therapy: results of a prospective, multicenter, double-blind, randomized, double-dummy, active-controlled trial. J Gastroenterol. 2012 May;47(5):540-52. doi: 10.1007/s00535-012-0541-z. Epub 2012 Mar 3. PMID 22388884
- [Derived] Geeratragool T, Kaosombatwattana U, Boonchote A, Chatthammanat S, Preechakawin N, Srichot J, Sudcharoen A, Sirisunhirun P, Termsinsuk P, Rugivarodom M, Limsrivilai J, Maneerattanaporn M, Pausawasdi N, Leelakusolvong S. Comparison of Vonoprazan Versus Intravenous Proton Pump Inhibitor for Prevention of High-Risk Peptic Ulcers Rebleeding After Successful Endoscopic Hemostasis: A Multicenter Randomized Noninferiority Trial. Gastroenterology. 2024 Sep;167(4):778-787.e3. doi: 10.1053/j.gastro.2024.03.036. Epub 2024 Apr 5. PMID 38582271